CLINICAL TRIAL: NCT02608671
Title: SKIN ADHESIVE TAPE COMPARED WITH CONTINUOUS SUTURE IN PERINEAL SKIN REPAIR AFTER EPISIOTOMY: RANDOMIZED TRIAL
Brief Title: Adhesive Tape in Episiotomy Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Lobna Ahmed Nabil (Unknown); Dr. Ahmed Sherif (Unknown); Dr. Mohamed Mahmoud El Sherbiny (Unknown); Prof. Mohamed Ashraf Mohamed Farouk Kortam (Unknown); Dr.Haitham Torky (Unknown)
Responsible Party: Principal Investigator, Ahmed Abass, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Adhesive tape&episiotomy
Record Dates: First submitted 2015-11-09; First posted 2015-11-20 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Episiotomy
Keywords: Episiotomy; continuous suture; Skin adhesive tape
MeSH Terms: interventions — Surgical Tape

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous skin suturing (No Intervention): will be subjected to skin repair after episiotomy with the currently traditional method for episiotomy repair by continuous absorbable subcuticular suture.
- Adhesive tape (Experimental): will be subjected to skin repair after episiotomy with skin adhesive tape.
  Interventions: Procedure: Skin adhesive tape

INTERVENTIONS:
Procedure: Skin adhesive tape
  Other Names: (® Steri-Strip
  Arms: Adhesive tape

SUMMARY:
This study will be undertaken to question the superiority of use skin adhesive tape (® Steri-Strip) closure system in wound healing over the traditional running absorbable subcuticular suture technique in perineal repair after episiotomy.

DETAILED DESCRIPTION:
Episiotomy is the most common operating procedure that most obstetricians will perform in their lifetime. Because it is so common and considered minor surgery, teaching students or interns the principles and techniques usually is left to the most junior of residents

The optimal method for episiotomy and perineal trauma repair following childbirth remains open to debate and a great cause of concern to doctors, midwives, and the public

Apparently, the ideal method for perineal repair should be quick, painless, easy to perform and preferably, without increase in pain and dyspareunia during the puerperium

This study will be undertaken to question the superiority of use skin adhesive tape (® Steri-Strip) closure system in wound healing over the traditional running absorbable subcuticular suture technique in perineal repair after episiotomy.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous.
* First and second degree perineal tear.
* Normal not instrumental vaginal delivery; spontaneous not induced.
* Patient willingness to randomize to episiotomy repair technique.

Exclusion Criteria:

* Previously existing local infections or lesions.
* Third and forth degrees perineal tear.
* Maternal diseases interfere with wound healing or causing excessive bleeding (coagulopathy, collagen disease, diabetes mellitus, known immunodeficiency, immunosuppressive treatment).
* Known hypersensitivity to adhesive materials
* Maternal unwillingness to undergo randomization.
* Participation in another intervention-trial with interference of intervention and/or outcome of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | During the procedure
  pain experience will be evaluated during the procedure,, 6 hours and 12 hours after the procedure by Wong-Baker faces pain rating scale .
  During the second visit 7-10 days after delivery; pain and patient satisfaction will be evaluated and recorded, data may be collected by phone for those may not be able to come back for the second visit.

SECONDARY OUTCOMES:
wound healing. | 10 days
  During the second visit 7-10 days after delivery; wound healing will be evaluated and recorded by Redness, Edema, Ecchymosis, Drainage, Approximation (REEDA), data may be collected by phone for those may not be able to come back for the second visit.
wound sepsis | 10 days
  During the second visit 7-10 days after delivery; wound sepsis will be evaluated and recorded by wound sepsis score, data may be collected by phone for those may not be able to come back for the second visit.
Postoperative pain | 2 hours after procedure
  pain experience will be evaluated 2 hours after the procedure by Wong-Baker faces pain rating scale .
Postoperative pain | 6 hours after procedure
  pain experience will be evaluated 6 hours after the procedure by Wong-Baker faces pain rating scale .
Postoperative pain | 12 hours after procedure
  pain experience will be evaluated 12 hours after the procedure by Wong-Baker faces pain rating scale .
Postoperative pain | 10 days after procedure
  pain experience will be evaluated by Wong-Baker faces pain rating scale .
timing of procedure | During the procedure
  timing of both procedures will be recorded and documented

REFERENCES:
- [Result] Feigenberg T, Maor-Sagie E, Zivi E, Abu-Dia M, Ben-Meir A, Sela HY, Ezra Y. Using adhesive glue to repair first degree perineal tears: a prospective randomized controlled trial. Biomed Res Int. 2014;2014:526590. doi: 10.1155/2014/526590. Epub 2014 Jun 26. PMID 25089271
- [Result] Ghosh A, Nanjappa M, Nagaraj V, Rajkumar GC. Comparison between stainless steel staples and silk sutures for primary closure of skin in patients undergoing neck dissection: A comparative clinical study. Contemp Clin Dent. 2015 Mar;6(Suppl 1):S51-5. doi: 10.4103/0976-237X.152938. PMID 25821376